CLINICAL TRIAL: NCT06000735
Title: Daily Blood Glucose Trends in Patients at Risk for Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Karol E. Watson, MD (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, Karol E. Watson, MD, Professor of Medicine, Cardiology, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-000975
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Stress; Blood Sugar; High; Cholesterol, Elevated; Diet Habit
MeSH Terms: conditions — Hyperglycemia; Hypercholesterolemia; Feeding Behavior | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: Pilot Study (uncontrolled)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 7-Day Continuous Glucose Monitoring with Abbott Freestyle Libre 2 (Experimental): All participants will go through the same intervention described above.
  Interventions: Device: 7-Day Continuous Glucose Monitoring with Abbott Freestyle Libre 2

INTERVENTIONS:
Device: 7-Day Continuous Glucose Monitoring with Abbott Freestyle Libre 2 — All participants will go through the same intervention described above

SUMMARY:
The goal of this study is to learn about the relationship between blood sugar, diet, stress, and metabolic parameters including waist circumference, body mass index (BMI), cholesterol levels and blood pressure in patients at risk for diabetes. The main questions it aims to answer are 1) are there trends in blood sugar responses after meals for patients at risk of developing diabetes? And 2) are there correlations between stress and fluctuations in blood sugar? During the first visit, participant's waist circumference, body composition, cholesterol, and resting blood pressure will be measured, and a continuous glucose monitor sensor will be placed on the participant's non-dominant arm. This sensor will be worn for seven days, and the participant will be asked to complete a daily food log during that time. Each participant will be asked to return to clinic after one week to return the continuous glucose monitor and daily food log.

DETAILED DESCRIPTION:
The relevance of diet, sleep, and stress and their metabolic consequences in cardiovascular risk is principal. Current improvements and developments in food labeling and personal self-tracking devices and applications (e.g. continuous glucose monitors [CGMs] and food logging apps), signal potential for better quantification of personal traits that could assist in defining personalized approaches for glycemic control. The objective of the proposed study is to evaluate daily glucose fluctuations and blood glucose time-in-range in relation to dietary intake and correlate excursions with metabolic risk factors in non-diabetic adults with one risk factor for diabetes mellitus. With the use of CGM technology to explore daily blood glucose trends in patients at risk for diabetes, the goal is to investigate relationships between blood glucose and metabolic parameters as well as sleep and stress factors.

The study will include two visits. During the first visit, the patient is explained the study details, their consent is obtained, their metabolic parameters measured, perceived stress scale questionnaire administered, and finally, the CGM is placed on them. The patient will be asked to return after one week to return the CGM reader, so the study team may collect the data.

ELIGIBILITY:
Inclusion Criteria (Must meet at least one of the following):

* Overweight and/or obese BMI classification, 25 to 35 kg/m2
* Fasting serum glucose ≥100 mg/dL and <126 mg/dL or HbA1c >5.7% and < 6.5%
* Family history of Type 2 DM
* History of hypertension, hypertriglyceridemia, heart disease, and/or stroke
* History of gestational diabetes

Exclusion Criteria:

* Any subject currently taking blood thinning medications such as Warfarin or Coumadin
* Any history of gastrointestinal disease or surgery except for appendectomy or cholecystectomy.
* History of gastrointestinal surgery, diabetes mellitus, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP >160mmHg, diastolic BP >95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, laxative abuse, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history.
* Pregnant or breastfeeding
* Currently uses tobacco products.
* Currently has an alcohol intake > 20 g ⁄ day;
* Currently has a coffee intake > 3 cups ⁄ day;
* Is unable or unwilling to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Blood glucose time-in-range (TIR) | 7 days
  The relationship between participants' TIR and cholesterol level, blood pressure, waist circumference, and perceived stress levels will be analyzed for any correlations.

CONTACTS AND LOCATIONS:
Overall Officials: Karol Watson, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Clinical Nutrition Clinic, 200 UCLA Medical Plaza, Suite 365-C, Los Angeles, California, United States